CLINICAL TRIAL: NCT03349255
Title: Phase 1, Open-label, Two Routes IV and Intra-hepatic Artery Dose-escalation Clinical Study to Evaluate the Safety and Efficacy of ET1402L1-CAR T- Cells in AFP Expressing Hepatocellular Carcinoma (HCC)
Brief Title: Clinical Study of ET1402L1-CAR T Cells in AFP Expressing Hepatocellular Carcinoma
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Will study new T-cell construct for the same indication
Sponsor: Aeon Therapeutics (Shanghai) Co., Ltd. (Industry)
Collaborators: Renmin Hospital of Wuhan University (Other); Eureka Therapeutics Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: ETCH17AFPCAR101
Record Dates: First submitted 2017-10-24; First posted 2017-11-21 (Actual); Last update posted 2019-07-01 (Actual); Status verified 2019-06

CONDITIONS: Hepatocellular Carcinoma; Liver Cancer; Liver Neoplasms; Metastatic Liver Cancer
Keywords: alpha-fetoprotein; AFP; HCC; CAR T cell therapy
MeSH Terms: conditions — Carcinoma, Hepatocellular; Liver Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- intravenous (i.v.) arm (Experimental): autologous ET1402L1-CART cells administered by intravenous (IV) infusion
  Interventions: Biological: autologous ET1402L1-CART cells
- intra-hepatic artery (i.a.) arm (Experimental): autologous ET1402L1-CART cells administered by intra-hepatic artery (IA) infusion
  Interventions: Biological: autologous ET1402L1-CART cells

INTERVENTIONS:
Biological: autologous ET1402L1-CART cells — Autologous T cells transduced with lentivirus encoding an anti-AFP (ET1402L1)-CAR expression construct

SUMMARY:
Clinical study to evaluate safety and pharmacokinetics (primary objectives) and efficacy (secondary objective) of ET1402L1-CART-cells in patients with AFP+ HCC

DETAILED DESCRIPTION:
The molecular target for ET1402L1-CART is alpha fetoprotein (AFP), which is expressed on 60-80 percent of hepatocellular carcinoma (HCC). ET1402L1-CART is a second generation (CD28/CD3ζ) chimeric antigen receptor (CAR) engineered with a human single-chain variable antibody fragments (scFv) against the anti-HLA-A02/AFP complex. This clinical study evaluates the safety and pharmacokinetics of ET1402L1-CART-cells in patients with HCC who have no available curative therapeutic options and a poor overall prognosis.

Patients with lesion(s) localized in liver will be enrolled in the IA arm, with the ET1402L1-CART-cells administered via intrahepatic artery catheter. Patients with extrahepatic metastasis will be enrolled in the IV arm, with the ET1402L1-CART-cells administered through intravenous infusion.

ELIGIBILITY:
Inclusion Criteria:

* AFP-expressing HCC and serum AFP >100 ng/mL.
* Measurable disease as defined by: at least 1 liver lesion that can be accurately and serially measured in at least 1 dimension and for which the longest diameter is ≥ 20 mm.
* Molecular HLA class I typing confirms participant carries at least one HLA-A02 allele
* Child-Pugh score of A or B
* Life expectancy > 4 months
* Age at time of enrollment is ≥18 years of age.
* KPS ≥70%
* Adequate organ function as defined below:

  * A pretreatment measured creatinine clearance (absolute value) of ≥50 ml/minute.
  * Patients must have a serum direct bilirubin ≤2 x ULN, ALT and AST ≤5 times the institutional upper limits of normal.
  * Ejection Fraction measured by echocardiogram or MUGA >45% (evaluation done within 6 weeks of screening does not need to be repeated)
  * DLCO or FEV1 >45% predicted
* Absolute neutrophil count (ANC) ≥ 1500/mm3 (10^9/L)
* Platelet count ≥ 50,000/mm3 (10^9/L)
* Negative serum pregnancy test for women with childbearing potential
* Informed Consent/Assent: All subjects must have the ability to understand and the willingness to sign a written informed consent.

Exclusion criteria:

* Patients with decompensated cirrhosis: Child-Pugh Score C
* Patients with an organ transplantation history
* Patients with tumor infiltration in the portal vein, hepatic veins or inferior vena cava that completely blocks circulation in liver.
* Patients with dependence on corticosteroids
* Patients with active autoimmune diseases requiring systemic immunosuppressive therapy
* Patients who are currently receiving or received within past 30 days anti-cancer therapy, local treatments for liver tumors (radiotherapy, embolism, ablation) or liver surgery
* Patients currently receiving other investigational treatments (biotherapy, chemotherapy, or radiotherapy)
* Patients undergoing current treatment known to interfere with lymphodepleting chemotherapy (cyclophosphamide, etc.).
* Participants with other active malignancies (except non-melanoma skin cancer and cervical cancer) within two years. Patients with a history of successfully-treated tumors with no sign of recurrence in the last two years may be enrolled.
* Patients with other uncontrolled diseases, such as active infections:

  * Acute or chronic active hepatitis B or hepatitis C.
  * HIV-infection
* Women who are pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2017-10-06 (Actual); Primary Completion 2019-01-10 (Actual); Study Completion 2019-01-10 (Actual)

PRIMARY OUTCOMES:
Number of patients with dose-limiting toxicity | 28 days up to 2 years
  A dose limiting toxicity is defined as any toxicity that is considered to be primarily related to the ET1402L1-CART-cells, which is irreversible, or life threatening or CTCAE Grade 3-5. Assessed at all visits.
Toxicity profile of ET1402L1-CART-cell treatment | 28 days up to 2 years
  Frequency of treatment-related adverse events that occurred at any time from the first day of infusion that are "possibly", "likely", or "definitely" related to the study, including infusion related toxicity and ET1402L1-CART T cells related toxicity. Include but not limited to: Fever, chills, nausea, vomiting, jaundice and other gastrointestinal symptoms; Fatigue, hypotension, respiratory distress; Tumor lysis syndrome; Cytokine release syndrome; Neutropenia, thrombocytopenia; Liver and kidney dysfunction. Assessed at all visits.

SECONDARY OUTCOMES:
Rate of disease response by RECIST in the liver | 2 years
  Response rates will be estimated as the percent of patients with objective response (OR), complete remission (CR), partial response (PR), stable disease (SD), no response (NR), overall survival (OS).
Rate of disease response by RECIST at non-liver sites | 2 years
  Response rates will be estimated as the percent of patients with objective response (OR), complete remission (CR), partial response (PR), stable disease (SD), no response (NR), overall survival (OS).
Anti-tumor responses | 4 months, 1 year, 2 years
  Progression free survival (PFS) and Median survival (MS) at 4 months, 1 year, 2 years
AFP serum levels | 2 years
  Percent change compared to the baseline
CART cell engraftment | 2 years
  Number and % of ET1402L1-CART cells in peripheral blood will be presented as Time to peak, Time to baseline level and the overall exposure will be presented as area under curve (AUC).
AFP expression in tumors | 4-8 weeks
  Percent of AFP-positive cells in randomly selected fields in tumor biopsies
Tmax of serum cytokine levels | 24 weeks
  Increases or decreases in the amount of cytokine produced compared to baseline at time points measured up to 24 weeks since dosing. Cytokines as measured by Bio-Plex Multiplex Immuoassays will be presented as time to peak level.
Time to baseline for serum cytokine levels | 24 weeks
  Increases or decreases in the amount of cytokine produced compared to baseline at time points measured up to 24 weeks since dosing. Cytokines as measured by Bio-Plex Multiplex Immuoassays will be presented as Time to baseline.
AUC of serum cytokine levels | 24 weeks
  Increases or decreases in the amount of cytokine produced compared to baseline at time points measured up to 24 weeks since dosing. Cytokines as measured by Bio-Plex Multiplex Immuoassays will be presented as area under curve (AUC).

CONTACTS AND LOCATIONS:
Overall Officials: Qibin Song, M.D./Ph.D., Principal Investigator — Renmin Hospital of Wuhan University
Locations (1):
- Renmin Hospital of Wuhan University, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: Undecided